CLINICAL TRIAL: NCT03110367
Title: Reframe the Pain: A Parent-Led Intervention to Alter Children's Memories for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Melanie Noel, Assistant Professor, University of Calgary, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB17-0426
Record Dates: First submitted 2017-03-18; First posted 2017-04-12 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Psychology; Pain; Stress; Behavior; Coping; Emotion, Expressed
MeSH Terms: conditions — Pain; Behavior

STUDY DESIGN:
Intervention Model Description: Participants will include 90 youth scheduled for a pectus repair or a spinal fusion surgery, surgeries associated with high levels of post-surgical pain, and their parents. They will be recruited at the Alberta Children's Hospital. The timelines and measures to be administered to parents and children are listed below. The timelines will include a baseline assessment (1-3 weeks pre-op), in hospital assessment for several days, 1-2 weeks post-op (acute recovery phase), the 2-4 week post-op clinic visit (memory reframing intervention) and 6 weeks post-op.
  Participants will be randomized into three groups:
  1. Attention Control Group
  2. Normal Reminiscing
  3. Intervention Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Reframing Intervention (Active Comparator): Participants will be randomized into this group:
  - Memory reframe with parent facilitated by researcher:
  Parents and youth in the intervention group will receive instructions about adaptive ways of reminiscing about the in-hospital and post-surgery periods. The intervention will draw from existing narrative-based interventions that have taught parents to reminisce with their children about past negative events in more elaborative and emotion-rich ways.
  Interventions: Behavioral: Pain Reframing Intervention
- Attention Control Group (Sham Comparator): Participants will include 90 youth scheduled for a pectus repair or a spinal fusion surgery, surgeries associated with high levels of post-surgical pain, and their parents. They will be recruited at the Alberta Children's Hospital. The timelines and measures to be administered to parents and children are listed below. The timelines will include a baseline assessment (1-3 weeks pre-op), in hospital assessment for several days, 1-2 weeks post-op (acute recovery phase), the 2-4 week post-op clinic visit (memory reframing intervention) and 6 weeks post-op.
  Participants will be randomized into this group:
  - Attention control (watch video [Planet Earth] for same amount of time): Parents and youth in the attention control group will watch a neutral 20-minute video that is not related to surgery (Planet Earth). Importantly, they will not talk about pain or the past surgery experience.
  Interventions: Behavioral: Attention Control Group
- Normal Reminiscing (No Intervention): Participants will include 90 youth scheduled for a pectus repair or a spinal fusion surgery, surgeries associated with high levels of post-surgical pain, and their parents. They will be recruited at the Alberta Children's Hospital. The timelines and measures to be administered to parents and children are listed below. The timelines will include a baseline assessment (1-3 weeks pre-op), in hospital assessment for several days, 1-2 weeks post-op (acute recovery phase), the 2-4 week post-op clinic visit (memory reframing intervention) and 6 weeks post-op.
  Participants will be randomized into this group:
  - Normal Reminiscing: Parents and youth in the normal reminiscing group will be instructed to reminisce with their children about the in-hospital and post-surgery periods as they normally would.

INTERVENTIONS:
Behavioral: Pain Reframing Intervention — Parents and youth in the intervention group will receive instructions about adaptive ways of reminiscing about the in-hospital and post-surgery periods. The intervention will draw from existing narrative-based interventions that have taught parents to reminisce with their children about past negative events in more elaborative and emotion-rich ways (e.g., using more open-ended questions, to follow in on children's answers by providing new details about the event, to talk more about emotions, and to praise children's answers).
  Arms: Pain Reframing Intervention
Behavioral: Attention Control Group — Parents and youth in the attention control group will watch a neutral 20-minute video that is not related to surgery (Planet Earth). Importantly, they will not talk about pain or the past surgery experience.
  Arms: Attention Control Group

SUMMARY:
Pain is a common experience in youth and influences youth long after the painful situations are over. Youth memory of pain after surgery can affect painful experiences in the future. Negative memories and feelings of pain, like remembering more pain than the actual level of pain experienced are linked to anxiety for future surgery. Research has found that children's memories of pain is linked to anxiety, pain-related fear, and confidence. Children's memories for pain can be altered after a visit to the hospital, but only a couple of studies have look at this.

The study will be one of the first to look at how well a parent-led memory reframing intervention to reduce youth's negative memories of surgery. We want to look at how a parent-led memory reframing session on youth's post-surgical pain memory.

The study will include 90 youth who have a chest wall surgery or a spinal fusion surgery at the Alberta Children's Hospital. They will be recruited at the Alberta Children's Hospital. There will be pain tests in the form of surveys 1-3 weeks before surgery, pain monitoring in the hospital for a couple of days, pain monitoring 1-2 weeks after surgery, a clinic visit 2-4 weeks after surgery for a memory reframing session, and pain monitoring 6 weeks after surgery in the form of a telephone interview.

DETAILED DESCRIPTION:
Background:

Children's pain memories are a powerful mechanism underlying subsequent pain experiences. Pain is ubiquitous in childhood. Healthy children who are compliant with medical care undergo up to 20 painful procedures by the age of 5. Moreover, millions of children undergo surgery (e.g., tonsillectomies) each year, which is commonly linked to pain and distress. Pain from, and fear of, medical experiences are neither short lasting or benign. Poorly managed pain can result in negatively biased pain memories, fears, and for some children, phobias that persist into adulthood. We have demonstrated that children's pain memories are a more important predictor of subsequent pain than their initial experience of pain itself. Indeed, children's pain memories fully mediated the relation between an initial and a subsequent laboratory pain experience. Our most recent data indicates that children's pain memories 2 months after surgery predict higher levels of post-surgical pain 4-6 months later.

Child and parent factors predict children's pain memory development. Existing research has implicated a number of factors in the development of negatively biased memories in children. Child sleep and language abilities have been shown to influence memory development following stressful and painful events. Children who are more anxious and who experience greater pain are more likely to develop negatively biased pain memories, which then leads to greater fear and pain at subsequent pain experiences. Parents and adolescents who think in more catastrophic ways about child pain prior to surgery tend to develop more negatively biased pain memories months later. Parent and child anxiety are thought to lead to memory biases because of the ways in which parents and children talk about pain following painful events. However, the influence of parent-child language-based interactions on pain memories has not been demonstrated.

The influence of parents on children's pain memories is greatest in early childhood. To guide future research on children's pain memory development, I published a conceptual developmental framework in the journal PAIN11 outlining the cognitive and social factors that are thought to influence children's pain memory development. Of particular importance is early childhood (ages 4-7 years) when children are most susceptible to memory biases due to suggestibility effects. It is also during this time that parents are most influential in shaping children's cognitions, emotions, and behaviors. Our model posits that the socio-linguistic context (e.g. parent-child narratives about pain) in which pain memories develop is most important in early childhood and sets the stage for future pain experiences.

Parent-child reminiscing influences children's memory development. Although surprisingly understudied in the field of pediatric pain, parent-child language-based interactions about past negative events, play a powerful role in how autobiographical memories of those events are subsequently retrieved and reframed. Parent-child narrative style also influences children's coping and psychological functioning. Young children whose parents are topic-extending and elaborative (e.g., who ask open-ended questions to pull for richer, more detailed accounts of the past) and who use emotional language, have children who are more accurate and detailed in recalling their pasts, which is adaptive. Similarly, our recent data provides strong evidence that parents who reminisce with their children about a recent surgery using a particular style (i.e., more elaborative, less topic-switching) and content (less content about pain, fear, medical procedures; more explanations) have children who later remember pain a more accurate/positively biased way.

Memory reframing interventions lead to children remembering pain in more accurate/positively-biased ways. To date, there have been three trials of memory reframing interventions, all of which were administered by a researcher to children undergoing needle procedures (vaccine injections, dental anesthetic injections, lumbar punctures) within 15 minutes. Our recent systematic review revealed that these interventions were efficacious in altering children's memories of pain to be more accurate/positively biased. Emphasizing and rehearsing positive aspects of a pain memory have also been shown to lead to an enhanced ability of children to forget its negative aspects. However, research has not yet implemented parent-led memory reframing interventions for children's pain; however, we have argued that parents are potentially the most powerful and accessible agents of change. Indeed, our recent data provides strong evidence that the language parents use when reminiscing with children following tonsillectomies influences children's pain memory biases.

Recent data from our lab provides compelling evidence that parents who reminisce with their children about surgery using a particular style (e.g., more elaborative, less topic-switching) and content (e.g., less content about pain, fear, medical procedures; more explanations) have children who later remember post-surgical pain a more accurate and positively biased way. Parental reminiscing style and content have been effectively targeted in interventions to improve children's memory development, albeit, not yet in the context of pain.To date, research has not examined if memory reframing techniques implemented by parents can alter children's recall of post-surgical pain. Thus, the goal of this research is to conduct a pilot study to examine the preliminary efficacy, feasibility, and acceptability of a brief parent-led memory reframing intervention following pediatric surgery to foster more adaptive (i.e., less negatively biased) pain memories. The intervention will draw from our recent data and extant memory reframing and narrative-based intervention techniques to promote more accurate/positive pain memories by teaching parents more adaptive styles of reminiscing with their children about a past surgery. We will accomplish our aims by extending our existing program of research on post-surgical pain memory development of children (aged 4-7 years) and randomly assigning parents to receive a memory reframing intervention or attention control following surgery and subsequently assessing children's memories for pain.

Study aims and hypotheses:

Aim 1.) To examine the preliminary efficacy, feasibility, and acceptability of a parent-led memory reframing intervention on children's post-surgical pain memories. Hypothesis 1.) Children in the intervention group will go on to recall post-surgical pain in a more accurate or positively biased way as compared to the control group who will remember pain in a more negatively biased way. The intervention will be judged by parents to be feasible and acceptable.

Aim 2.) To examine the influence of baseline individual child and parent characteristics on children's pain memories. Hypothesis 2.) Children who are more anxious, less self-efficacious, have worse sleep quality, and whose parents are more anxious and catastrophize more about child pain prior to surgery will subsequently remember pain in a more negatively biased way.

This study will be the first to develop and pilot test a brief, parent-led intervention aimed at changing the way children recall their pain after surgery, thereby extending memory-reframing techniques to the post-surgical pain context. Given the integral role of pain memories in shaping future pain experiences and the need for interventions in the pediatric surgery context, this study has great potential to contribute an accessible and feasible post-surgical pediatric pain management intervention and foster more adaptive pain trajectories and medical experiences in childhood.

Methods:

Sample:

Participants will include 90 adolescents scheduled for a pectus repair or spinal fusion, surgeries associated with high levels of post-surgical pain,2 and their parents. They will be recruited at the Alberta Children's Hospital (ACH). We will use a recruitment strategy that is consistent with our studies with clinical samples. Specifically, the recruitment pool will be generated as follows: 1) clinic staff will identify the patients scheduled for pectus repair or spinal fusion surgeries; 2) upon booking of the pre-op clinic visit, the admin staff will obtain permission to contact for research purposes from parents along with contact details; 3) clinic staff will pass on the contact information to the research study team via a secure electronic transfer; 4) the study staff will contact eligible families and screen interested parents and youth for eligibility and address any questions they might have and then set up a time to conduct a consent conference call with parent and child. This consent call will involve a discussion with the parent and child who will participate in the study and a researcher. The researcher will explain the information included in the consent form and provide the opportunity for potential participants to ask questions and clarify understanding. At this time, we will also clearly outline our limits to confidentiality regarding disclosure of abuse, neglect, suicidal ideation and intent, and potential to a minor. These are described on the consent form; however, the consent conference is an excellent opportunity to reiterate and clarify these procedures and issues. For this consent conference, a researcher will email these forms to participants (using REDCap, a secure online web-based application) who can complete them on a computer device. To increase participation, we will also distribute the posters (see Recruitment Poster) within ACH, so that potential participants will have the opportunity to contact us directly to indicate interest in the study. Screening for eligibility and consent procedures will be as described above.

Procedure:

One week before surgery, youth will complete measures of pain, sleep (Adolescent Sleep Wake Scale; ASWS), pain catastrophizing (PCS - Child version), anxiety and depression symptoms (PROMIS-25), quality of life (PedsQL), PTSD symptoms (CPSS-5), sensitivity to pain traumatization (SPTS-Child version), self-efficacy about pain, expectancies about pain and pain-related fear (Numerical Rating Scales; NRS). Parents will complete measures of sleep (Pittsburgh Sleep Quality Index), pain catastrophizing (PCS-Parent version), measures of anxiety, depression and PTSD symptoms (PROMIS-29 and PCL-5), sensitivity to pain traumatization (SPTS-Parent version), self-efficacy about pain, parent responses to child pain (ARCS), expectancies about pain and pain-related fear (NRS), a socio-demographic survey (parent education, child age, household income), preparation that they/their child received about the surgery and what this entailed (e.g., coping skills, pain management), and family history of surgeries.

On the day of surgery and every day after the surgery (until discharge), both youth and parents will report pain characteristics (pain intensity [NRS], pain-related fear [NRS], pain interference [PROMIS], pain unpleasantness [a Likert scale], pain catastrophizing [state]), state anxiety (NRS), overall affect (NRS), and sleep quality (NRS). Parents will also complete a measure of parent responses to child pain (ARCS). Information regarding analgesic and anesthetic agents administered on the day of surgery will be collected via medical chart review.

At 2-weeks post-surgery, parents and youth will complete the baseline assessment measures.

At 4-weeks post-surgery following their clinic visit, parent-child dyads will be randomized into three groups: an attention control group, a normal reminiscing group, and an intervention group. Randomization will be conducted by an external statistician using a computer random number generator. Allocation concealment will be achieved using sequentially numbered, opaque, and sealed envelopes. Group allocation will be revealed by a researcher at the outset of the lab visit.

Attention Control Group: Parents and youth in the attention control group will watch a neutral 20-minute video that is not related to surgery (Planet Earth). Importantly, they will not talk about pain or the past surgery experience.

Normal Reminiscing: Parents and youth in the normal reminiscing group will be instructed to reminisce with their children about the in-hospital and post-surgery periods as they normally would.

Intervention Group: Parents and youth in the intervention group will receive instructions about adaptive ways of reminiscing about the in-hospital and post-surgery periods. The intervention will draw from existing narrative-based interventions that have taught parents to reminisce with their children about past negative events in more elaborative and emotion-rich ways (e.g., using more open-ended questions, to follow in on children's answers by providing new details about the event, to talk more about emotions, and to praise children's answers). We will also include elements of past pain memory reframing interventions and findings from our recent data. Specifically, parents will be taught to reminisce with their children about the in-hospital and post-surgery periods by providing more explanations for events, using less utterances about pain, fear, and medical procedures, emphasizing positive aspects of the child's surgery memory (e.g., when children used coping methods such as deep breathing, when they got a treat), and enhancing children's self-efficacy regarding their ability to cope with pain. Researchers will also provide suggestions for specific questions and remarks to make while reminiscing. Parents, youth, and researchers will engage in brief role-plays to solidify the techniques, which will be followed by researcher feedback. After this training period, parents in the intervention group will be instructed to reminisce with their children about the in-hospital and post-surgery periods using the intervention strategies.

At 6-weeks post-surgery, youth and parent will complete a telephone pain memory interview to assess youth's recall of the in-hospital and post-surgery periods.Then, parents in the intervention group will complete a brief semi-structured telephone interview to assess feasibility and acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Youth between the age of 10 to 18
2. Youth who are scheduled to have a chest wall surgery or a spinal fusion surgery

Exclusion Criteria:

1. Youth with developmental disorders or who are being treated for cancer
2. Youth who have had a chest wall surgery or spinal fusion surgery before
3. Youth who are scheduled for other surgical procedures within 24 hours of the scheduled chest wall surgery or spinal fusion surgery
4. Youth who do not speak fluent English
5. Youth who have two non-fluent English speaking parents (one parent must be fluent in English to participate)
6. Youth who experience chronic pain

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Memory Biases | 4 weeks post-operative (for spinal instrumentation surgeries) - 6 weeks post operative (for pectus chest wall surgeries)
  Youth and parents will complete telephone memory interviews to assess their pain memories. Specifically, youth will be asked to remember the levels of sensory (pain intensity) and affective (unpleasantness, anxiety) pain experienced after the surgery. Parents will be asked to remember the levels of sensory (pain intensity) and affective (unpleasantness, anxiety) pain they think their children experienced after the surgery. At the beginning of the memory interviews, children and parents will be asked to freely recall anything that they can remember about the pain task. Telephone interviews to assess children's memory for pain have been effectively conducted with youth. Positively biased pain memories will be defined as recalled pain level that is less than the initial pain report. Accurate memories reflect no difference between recalled and experienced pain. Free recall will be coded for both content and tone.

SECONDARY OUTCOMES:
Sleep Quality - Child | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  The 10-item short-form of the Adolescent Sleep Wake Scale (ASWS) will be used to assess sleep quality in youth. The ASWS assesses sleep quality along 3 dimensions: Falling asleep and reinitiating sleep, returning to wakefulness, and going to bed. This measure has good reliability and validity in youth with chronic pain. Post-surgical sleep quality will be assessed using an NRS (0 = extremely poor sleep, 10 = extremely good sleep).
Sleep quality - Parent | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  Parent quality of sleep over the last month will be assessed using a well-validated and widely used Pittsburgh Sleep Quality Index (PSQI). Nineteen items comprise seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The component scores are summed to yields the global score. The PSQI is reliable and valid.
Pain Intensity | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries), telephone interview (6 weeks post operative)
  Youth will rate their pain intensity an 11-point NRS (0 - no pain; 10 - worst pain possible). NRSs are a valid and reliable tool to assess pain intensity in youth.35,36 Average pain scores will be computed for each assessment period. The NRS will be included in the memory interviews but framed in terms of recall of pain. Parents will use the same scale to assess their child's pain.
Pain characteristics, unpleasantness, and interference. | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  The 7-item Pain Questionnaire assesses pain frequency, location, duration, intensity, distress, and interference. The pain unpleasantness item is rated on a 5-point Likert scale assessing how much pain bothered the child. Pain interference will be measured using the pain interference subscale of the PROMIS-25 Profile. The subscale's four items are rated on a 5-point Likert scale and assess the extent of everyday impairment due to pain. The scale has excellent psychometric properties and has been used in youth with chronic pain.
Pain-related anxiety. | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries), telephone interview (6 weeks post operative)
  Anticipatory and experienced pain-related anxiety related to the pre- and post-surgical pain will be assessed using an 11-point NRS (0 = "not anxious/nervous", 10 = "extremely nervous or anxious") (child and parent report). Similar scales have been used in previous research on children's pain. This measure will be included in the memory interviews but framed in terms of recall.
Post-traumatic stress disorder symptoms - Child | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  The 27-item Child PTSD Symptom Scale (CPSS-V) will be used to assess PTSD symptoms according to DSM-5 diagnostic criteria. Twenty symptoms are rated on a 4-point Likert scale; 7 impairment items are rated as present or absent. Total and cluster specific symptom scores and impairment scores are yielded. The CPSS-5 is based on the CPSS-4, which has excellent psychometric properties. We used this scale in our pilot research.
Anxiety and depressive symptoms - child | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  Youth anxiety and depressive symptoms will be assessed using the PROMIS-25 Pediatric profile, one of the Pediatric Profile instruments developed by the National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS). Twenty-five items of the measure assess anxiety and depressive symptoms, physical function mobility, fatigue, peer relationships, pain interference, and pain intensity on a 5-point Likert scales.
Physical and psychosocial functioning. | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  The 15-item Pediatric Quality of Life Scale (PedsQL) assesses health-related physical, emotional, social, and school functioning using a 5-point Likert scale. The PedsQL is widely used in illness and healthy samples and has excellent psychometric properties.
Sensitivity to pain traumatization (Child version). | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  This 12-item Sensitivity to Pain Traumatization Scale - Child version (SPTS-C) has been developed based on the adult version of the scale (SPTS) to assess anxiety-related reactions to pain that are similar to symptoms of posttraumatic stress disorder. The items are rated on a 5-point Likert scale, a higher total score indicates a higher level of sensitivity to pain traumatization.
Catastrophic thinking about pain - Trait (Child) | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  Catastrophizing Scale-Child Version (PCS-C) is a 13-item measure assessing children's catastrophic thoughts and feelings about their pain. Items are rated on a 5-point Likert scale. Among youth with pain, the PCS-C has good validity and reliability.
Catastrophic thinking about pain - State (Child version). | assessment will take place on day 1 post-operative (day after surgical procedure), day 2 post-operative, day 3 post-operative, day 4 post-operative, day 5 post-operative (if applicable - not yet discharged)
  During first days after surgery (until discharge) youth will be asked to rate six statements on an 11-point NRS ("not at all" and "a lot" anchors). The statements correspond to the three PCS-C subscales, i.e., rumination, magnification, helplessness, and adapted from the PCS-C.
Parent responses to child pain. | assessment will take place on day 1 post-operative (day after surgical procedure), day 2 post-operative, day 3 post-operative, day 4 post-operative, day 5 post-operative (if applicable - not yet discharged)
  The 26-item Adult Responses to Children's Symptoms (ARCS) with a pain-specific stem will be used to assess parents' responses to child pain complaints. Frequency of behaviours is rated on a 5-point Likert scale. This measure is both valid and reliable. Protect scale of the ARCS will be completed by parents every day post-surgery up to discharge.
Background variables collected at baseline - child age | collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Pain characteristics, unpleasantness, and interference (Subscale) | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  The subscale's four items are rated on a 5-point Likert scale and assess the extent of everyday impairment due to pain. The scale has excellent psychometric properties and has been used in youth with chronic pain.
Post-traumatic stress disorder symptoms - Parent | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  Parents' PTSD symptoms will be assessed using the 20-item PTSD Checklist for DSM-5 (PCL-5) with an extended Criterion A and a Life Events Checklist. Response options are rated on a 4-point Likert scale. Total symptom severity and cluster-specific scores are obtained. The measure is valid and reliable. We used this measure in our pilot research on PTSD and chronic pain in youth and parents.
Sensitivity to pain traumatization (Parent version). | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  The 12-item Sensitivity to Pain Traumatization Scale - Parent version (SPTS-P) has been developed based on the adult version of the scale (SPTS) to assess parental anxiety-related reactions to pain in their children that are similar to symptoms of posttraumatic stress disorder. The items are rated on a 5-point Likert scale, a higher total score indicates a higher level of sensitivity to pain traumatization.
Catastrophic thinking about pain - Trait (Parent) | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  The Pain Catastrophizing Scale-Parent Version (PCS-P) is a 13-item self-report measure assessing catastrophic thoughts and feelings that parents may have when their child experiences pain. Items on the PCS-P are rated on a 5-point Likert scale. The PCS-P is both valid and reliable among parents of youth with and without chronic pain.
Catastrophic thinking about pain - State (Parent version). | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  Parents will be asked to rate six statements on an 11-point NRS ("not at all" and "a lot" anchors). The statements correspond to the three PCS-P subscales, i.e., rumination, magnification, helplessness, and adapted from the PCS-P.
Anxiety and depressive symptoms - Parent | At baseline, in hospital assessment (1-5 days after surgery), 1 week post surgery (for spinal instrumentation surgeries) - 2 weeks post surgery (for pectus chest wall surgeries)
  Parents' anxiety and depressive symptoms will be assessed using the PROMIS-29 profile, an adult version of PROMIS-25 profile assessing the same areas of functioning.
Background variables collected at baseline - parent age | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variable collected at baseline - parent sex | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - child sex | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - child school status | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - parent race | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - child race | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - parent marital status | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - child marital status | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - child education | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - parent education | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.
Background variables collected at baseline - family income | Collected at baseline
  Parents will complete a questionnaire reporting on demographic characteristics of themselves and their children including: age, sex, school status (e.g., attendance, specialized programming such as an individualized program plan [IPP]), race, marital status, education, and family income. We will request a copy of an IPP from those participants who have it. It will be used to further understand contextual support systems that is available to youth.

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavlova M, Lund T, Sun J, Katz J, Brindle M, Noel M. A memory-reframing intervention to reduce pain in youth undergoing major surgery: Pilot randomized controlled trial of feasibility and acceptability. Can J Pain. 2022 Jun 9;6(2):152-165. doi: 10.1080/24740527.2022.2058919. eCollection 2022. PMID 35711298